CLINICAL TRIAL: NCT05823454
Title: Consciousness-specific Brain Network Connection of Propofol Sedation and Prolonged Disorders of Consciousness Based on Electroencephalogram and Event-related Potential
Brief Title: Consciousness-specific Brain Network Connection of Propofol Sedation and Prolonged Disorders of Consciousness
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Other Study IDs: ywn20220929
Record Dates: First submitted 2023-03-05; First posted 2023-04-21 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Consciousness Disorder
Keywords: Prolonged Disorders of Consciousness; Propofol; Brain Functional connectivity; Electroencephalography
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Propofol: Intravenous infusion
  Interventions: Drug: Different drug dosage
- Dexmedetomidine: Intravenous infusion
  Interventions: Drug: Different drug dosage
- Esketamine: Intravenous infusion
  Interventions: Drug: Different drug dosage
- Sevoflurane: Inhalation anesthesia
  Interventions: Drug: Different drug dosage
- Remifentanil: Intravenous infusion
  Interventions: Drug: Different drug dosage

INTERVENTIONS:
Drug: Different drug dosage — Choice of Anesthesia

SUMMARY:
Consciousness-specific Brain Network Connection of Propofol Sedation and Prolonged Disorders of Consciousness based on Electroencephalography and Auditory Event-related Potentials

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years old, native Chinese speaker, dextromanuality;
* Chronic disorder of consciousness;
* Spinal cord electrical stimulator implantation under general anesthesia;
* Signed informed consent.

Exclusion Criteria:

* Continuous sedation was administered within 72 hours prior to the study;
* Open head injury, parenchymatectomy and other damage of brain structural integrity;
* The intracranial compliance decreased due to hydrocephalus and swelling;
* Known hearing impairment;
* Airway stenosis and various causes of severe ventilation or ventilation dysfunction;
* Known or suspected cardiac dysfunction;
* Allergic to intravenous general anesthetics;
* Associated with other mental or neurological diseases;
* Other reasons are not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with chronic disorders of consciousness
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
EEG Spectral Characteristics | During the trial(up to 3 hours for each subject)
  Characteristics of EEG power spectrum(for 1-30 Hz) in patients with chronic consciousness disorder under different doses of drugs

SECONDARY OUTCOMES:
Cortical Connectivity | During the trial(up to 3 hours for each subject)
  Characteristics of the weighted phase lag index in patients with chronic consciousness
Derived quantitative indicators | During the trial(up to 3 hours for each subject)
  Characteristics of EEG derived quantitative indicators with chronic consciousness disorder during anesthesia recovery
Characteristics of sleep | During the trial(up to 24 hours for each subject)
  Characteristics of sleep cycle in patients with chronic disorders of consciousness
Dynamic Patterns of Cortical Connectivity | During the trial(up to 3 hours for each subject)
  The time-frequency characteristics of the weighted phase lag index in patients with chronic disorders of consciousness
Rate of patients recovered consciousness after surgery | During the trial(through study completion, 180 days)
  Rate of patients recovered consciousness 30 days, 90 days, 180 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No